CLINICAL TRIAL: NCT00821249
Title: A Study of ARRY-520 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-520-212
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Multiple Myeloma; Plasma Cell Leukemia
Keywords: plasma cell dyscrasia; plasmacytoma; kinesin spindle protein; anti-mitotic
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell; Paraproteinemias; Plasmacytoma | interventions — filanesib; Filgrastim; Granulocyte Colony-Stimulating Factor; Injections, Subcutaneous; Dexamethasone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARRY-520 (Experimental)
  Interventions: Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous
- ARRY-520 + G-CSF support (Experimental)
  Interventions: Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous; Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous
- ARRY-520 + dexamethasone + G-CSF support (Experimental)
  Interventions: Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous; Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous; Drug: Dexamethasone, steroid; oral

INTERVENTIONS:
Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous — Part 1: multiple dose, escalating; Part 2: multiple dose, single schedule; Part 3: multiple dose, single schedule.
Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous — Part 1: standard of care; Part 2: standard of care; Part 3: standard of care.
  Arms: ARRY-520 + G-CSF support; ARRY-520 + dexamethasone + G-CSF support
Drug: Dexamethasone, steroid; oral — Part 3: standard of care.
  Arms: ARRY-520 + dexamethasone + G-CSF support

SUMMARY:
This is a 2-phase study during which patients with relapsed or refractory multiple myeloma (MM) or plasma cell leukemia (PCL), who have already received at least two previous treatments, will receive investigational study drug ARRY-520.

The study has 3 parts. In the first part of the study, Phase 1, patients will receive increasing doses of study drug, with or without granulocyte-colony stimulating factor (G-CSF) support, in order to achieve the highest dose possible that will not cause unacceptable side effects. Approximately 30 patients from the US will be enrolled in Part 1 (Active, not recruiting).

In the second part of the study, Phase 2, patients will receive the best dose of study drug determined from the first part of the study and will be followed to evaluate what side effects the study drug causes and what effectiveness it has, if any, in treating the cancer. Approximately 30 patients from the US will be enrolled in Part 2 (Active, not recruiting).

In the third part of the study, Phase 2 with Dexamethasone, patients will receive the best dose of the study drug determined from the first part of the study, in combination with dexamethasone, and will be followed to evaluate what side effects the combination causes and what effectiveness the combination has, if any, in treating the cancer. Approximately 50 patients from the US will be enrolled in Part 3 (Active, not recruiting).

ELIGIBILITY:
Key Inclusion Criteria (Part 3):

* Patients should have received at least two prior treatment regimens.
* Confirmed refractory MM (measurable disease) or PCL. Patients must be refractory to treatment with both lenalidomide/dexamethasone and bortezomib/dexamethasone (or to treatment with bortezomib/lenalidomide/dexamethasone), defined as documented progressive disease on therapy or within 60 days of completing treatment with these regimens.
* Previously received adequate alkylator therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Adequate hematology laboratory values without transfusion support within 2 weeks of screening.
* Adequate liver and renal function.
* Additional criteria exist.

Key Exclusion Criteria (Part 3):

* Primary amyloidosis.
* Concomitant malignancies or previous malignancies with less than a 3-year disease free interval at the time of enrollment (patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or Stage A low grade prostate cancer may enroll irrespective of the time of diagnosis).
* Autologous or allogeneic stem cell or bone marrow transplant within 3 months prior to first dose of study drug.
* Cytotoxic therapy or monoclonal antibodies within 21 days prior to first dose of study drug.
* Radiotherapy within 21 days prior to first dose of study drug (if the radiation portal covered ≤ 5% of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy).
* Corticosteroid doses > 10 mg/day of prednisone or equivalent within 2 weeks prior to first dose of study drug.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis B and/or active hepatitis C.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of study drug, with and without G-CSF. | Part 1
Assess the efficacy of the study drug, with and without dexamethasone, in terms of response rate. | Part 2 and Part 3
Characterize the safety profile of the study drug in combination with dexamethasone in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 3

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of the study drug. | Part 1
Assess the efficacy of the study drug in terms of response rate, duration of response, progression-free survival, treatment-free survival and time to next treatment. | Part 1
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 2
Assess the efficacy of the study drug, with and without dexamethasone, in terms of duration of response, progression-free survival, treatment-free survival, time to next treatment and overall survival. | Part 2 and Part 3
Explore potential biomarkers for pharmacodynamics (PD) and for patient selection. | Part 1, Part 2 and Part 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Shah JJ, Kaufman JL, Zonder JA, Cohen AD, Bensinger WI, Hilder BW, Rush SA, Walker DH, Tunquist BJ, Litwiler KS, Ptaszynski M, Orlowski RZ, Lonial S. A Phase 1 and 2 study of Filanesib alone and in combination with low-dose dexamethasone in relapsed/refractory multiple myeloma. Cancer. 2017 Dec 1;123(23):4617-4630. doi: 10.1002/cncr.30892. Epub 2017 Aug 17. PMID 28817190